CLINICAL TRIAL: NCT07348016
Title: Safety and Efficacy of Platelet-Rich Plasma Combined With Compound Betamethasone in Arthroscopic Surgery for Rotator Cuff Injury With Shoulder Adhesion: A Prospective, Multicenter, Randomized Controlled Trial
Acronym: PRP+CB for RC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFY-2025-085; EFY-2025-085 (Other Grant/Funding Number: The Second Affiliated Hospital of Nanchang University)
Record Dates: First submitted 2025-12-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Injuries; Adhesions
Keywords: Platelet-Rich Plasma; Compound Betamethasone; Arthroscopy; Randomized Controlled Trial; Shoulder; Stiffness
MeSH Terms: conditions — Rotator Cuff Injuries; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The injection syringes will be prepared by a research pharmacist or designated staff member not involved in patient assessment. Both the experimental (PRP + Compound Betamethasone) and control (normal saline placebo) injections will be identical in appearance (color and volume). Participants, surgeons, postoperative care providers, and outcome assessors will all be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy Group (Experimental): Participants will receive arthroscopic rotator cuff repair and adhesion release, followed by an intra-articular injection of Liposomal Bupivacaine combined with Compound Betamethasone.
  Interventions: Drug: Liposomal Bupivacaine + Compound Betamethasone Injection
- Monotherapy (Control) Group (Active Comparator): Participants will receive arthroscopic rotator cuff repair and adhesion release, followed by an intra-articular injection of Compound Betamethasone alone.
  Interventions: Drug: Compound Betamethasone Injection

INTERVENTIONS:
Drug: Liposomal Bupivacaine + Compound Betamethasone Injection — Intra-articular injection of a mixture containing Liposomal Bupivacaine and Compound Betamethasone under arthroscopic guidance after standard surgical procedures.
  Arms: Combination Therapy Group
Drug: Compound Betamethasone Injection — Intra-articular injection of Compound Betamethasone alone under arthroscopic guidance after standard surgical procedures.
  Arms: Monotherapy (Control) Group

SUMMARY:
Background: Patients undergoing arthroscopic surgery for rotator cuff tears with shoulder adhesion often experience significant postoperative pain and stiffness. This study investigates whether adding a long-acting local anesthetic (Liposomal Bupivacaine) to a standard anti-inflammatory steroid injection (Compound Betamethasone) during surgery can improve outcomes.

Methods: This is a prospective, randomized, double-blind, controlled trial. Approximately 70 eligible adult patients will be randomly assigned to one of two groups: (1) the Combination Group, receiving an intra-articular injection of Liposomal Bupivacaine plus Compound Betamethasone after surgery, or (2) the Control Group, receiving Compound Betamethasone alone. Patients and outcome assessors will not know the group assignment.

What participants will do: All participants will receive standard arthroscopic rotator cuff repair and adhesion release. They will be followed for 12 months after surgery, with assessments at multiple time points (from hours to months post-op) to measure pain levels, shoulder function, range of motion, and tendon healing via MRI.

Main Goals: The primary goal is to compare the improvement in UCLA shoulder scores between the two groups at 12 months. Secondary goals include comparing pain scores, other functional scores (Constant-Murley), joint mobility, MRI findings, and safety (complication rates).

DETAILED DESCRIPTION:
Study Design: A prospective, randomized, double-blind, parallel-group, active-controlled clinical trial conducted at The Second Affiliated Hospital of Nanchang University.

Participants & Sample Size: 70 patients (35 per group) with full-thickness rotator cuff tear and concomitant shoulder adhesion scheduled for arthroscopic repair. Sample size was calculated based on an expected difference in UCLA scores with 80% power and α=0.05, accounting for a 20% dropout rate.

Interventions:

Combination Therapy Group: After standard arthroscopic rotator cuff repair and capsular release, the shoulder joint will be injected with a mixture of Liposomal Bupivacaine and Compound Betamethasone under direct visualization.

Active Control Group: After the same surgical procedure, the joint will be injected with Compound Betamethasone alone.

Outcome Measures:

Primary: UCLA Shoulder Score (assessed pre-op, 3, 6, 12 months).

Secondary: Visual Analog Scale (VAS) for pain (assessed at 11 time points from pre-op to 12 months), Constant-Murley Shoulder Score, active range of motion (forward flexion, abduction), MRI evaluation of tendon healing using Signal-to-Noise Quotient (SNQ) of the supraspinatus tendon (distal and proximal), and incidence of complications (infection, re-tear, thrombosis, adhesion) within 12 months.

Statistics: Data will be analyzed using SPSS. Continuous variables will be compared using t-tests or non-parametric tests as appropriate. Categorical variables will be compared using Chi-square tests. A p-value <0.05 will be considered statistically significant.

Ethics & Registration: The study protocol will be submitted for approval to the Institutional Review Board of The Second Affiliated Hospital of Nanchang University. It will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines. This trial is registered on ClinicalTrials.gov.

Funding: Supported by the Internal Grant Program of The Second Affiliated Hospital of Nanchang University.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 70 years.

Clinical and MRI diagnosis of full-thickness rotator cuff tear.

Presence of shoulder stiffness/adhesion defined as passive range of motion less than 100° in forward flexion and/or less than 10° in external rotation (or according to your specific definition).

Scheduled for arthroscopic rotator cuff repair and capsular release.

Willing and able to provide written informed consent.

Willing to comply with all study procedures and follow-up visits.

Exclusion Criteria :

Massive, irreparable rotator cuff tear.

Severe glenohumeral osteoarthritis (Grade III or IV according to Samilson-Prieto classification).

History of shoulder infection, fracture, or previous surgery on the affected shoulder.

Known allergy or contraindication to betamethasone, local anesthetics, or components of PRP preparation.

Systemic inflammatory arthritis (e.g., rheumatoid arthritis).

Coagulation disorders or use of anticoagulants that cannot be safely suspended perioperatively.

Pregnancy or lactation.

Participation in another clinical trial within the past 3 months.

Any medical or psychiatric condition that, in the investigator's opinion, would compromise patient safety or compliance with the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Constant-Murley Shoulder Score | Baseline, 3 months, and 12 months postoperatively.
  The Constant-Murley score is a composite outcome measure assessing shoulder pain, activities of daily living, range of motion, and strength. Scores range from 0 to 100, with higher scores indicating better function.
Visual Analog Scale (VAS) Pain Score at Rest | Baseline, 3 months, and 12 months postoperatively.
  Pain intensity at rest measured on a 100-mm Visual Analog Scale, where 0 mm represents "no pain" and 100 mm represents "worst pain imaginable."

SECONDARY OUTCOMES:
Active Range of Motion (ROM) | Baseline, 3 months, and 12 months postoperatively.
  Measured in degrees for shoulder forward flexion, abduction, and external rotation using a goniometer
American Shoulder and Elbow Surgeons (ASES) Score | Baseline, 3 months, and 12 months postoperatively.
  A patient-reported outcome measure assessing pain and functional activities. Scores range from 0 to 100, with higher scores indicating better function.
MRI Assessment of Tendon Healing | 3 months and 12 months postoperatively.
  MRI Assessment of Tendon Healing
Incidence of Treatment-Related Adverse Events | From the time of surgery up to 12 months postoperatively.
  Number and severity of adverse events (e.g., infection, allergic reaction, abnormal bleeding, systemic effects) assessed as related to the study interventions (PRP and/or betamethasone injection).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No